CLINICAL TRIAL: NCT00319800
Title: A Phase II Study of Second-Line Therapy With Irinotecan or Gefitinib in Docetaxel Pretreated Patients With Non-Small Cell Lung Cancer: a New Treatment Strategy According to Clinical Predictors for Response
Brief Title: Second-Line Irinotecan or Gefitinib in Docetaxel Pretreated NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMO-LU-62
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Irinotecan

INTERVENTIONS:
Drug: Gefitinib
Drug: Irinotecan

SUMMARY:
To determine whether in docetaxel pretreated advanced NSCLC patients with favorable clinical parameter(s) gefitinib can produce different outcomes from patients without favorable clinical parameter treated with irinotecan.

DETAILED DESCRIPTION:
It has been suggested that some clinical parameters, including women, no smoking history and a histologic diagnosis of adenocarcinoma, are associated with favorable outcomes of gefitinib therapy. We will conduct a phase II study in docetaxel pretreated advanced NSCLC patients treated with gefitinib or irinotecan according to these clinical parameters in order to determine whether in patients with favorable clinical parameter(s) gefitinib will produce difference outcomes from patients without favorable clinical parameter treated with irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* aged 75 years or less
* histologically or cytologically confirmed non-small cell lung cancer
* advanced, metastatic or recurrent
* ECOG performance status 0 to 2
* one prior palliative chemotherapy including docetaxel
* measurable or evaluable indicator lesion(s)
* normal marrow, hepatic and renal function
* provision of written informed consent

Exclusion Criteria:

* active infection and/or severe comorbidities
* pregnant or breastfed women
* active CNS metastasis
* active bleeding in GI tract or elsewhere

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-02; Study Completion 2007-03

PRIMARY OUTCOMES:
Objective response rate
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Gachon University Gil Medical Center, Incheon, Korea
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea